CLINICAL TRIAL: NCT05720130
Title: Phase Ib/IIa Dose Escalation and Expansion Study of [²¹²Pb]Pb-ADVC001 in Metastatic Castration Resistant Prostate Cancer (TheraPb - Phase I/II Study).
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AdvanCell Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TheraPb-ADVC001
Record Dates: First submitted 2023-01-07; First posted 2023-02-09 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Prostate Cancer; Metastatic Castration-resistant Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- mCRPC (Experimental): Phase 1b Dose Escalation: Participants with PSMA-positive mCRPC who have had exposure to at least one ARPi and taxane-based chemotherapy (unless taxanes contraindicated or declined) at any time in the course of their disease.
  Phase 2a Dose Expansion:
  Group 1: Participants with PSMA-positive mCRPC who have had exposure to at least one ARPi at any time in the course of their disease and received taxane-based chemotherapy for the treatment of mCRPC.
  Group 2: Participants with PSMA-positive mCRPC who have had exposure to at least one ARPi at any time in the course of their disease and has not received a taxane for the treatment of mCRPC.
  Group 3: Participants with PSMA-positive mCRPC who have had exposure to at least one ARPi and to 177Lu-PSMA at any time in the course of their disease.
  Interventions: Drug: [²¹²Pb]Pb-ADVC001

INTERVENTIONS:
Drug: [²¹²Pb]Pb-ADVC001 — Ph1b Escalation
  Drug: [²¹²Pb]Pb-ADVC001administered intravenously per dose escalation scheme
  Dose Level 1
  - 60 MBq, 4 cycles every 6 weeks
  Dose Level 2a
  - 120 MBq, 4 to 6 cycles every 4 weeks
  Dose Level 2b
  - Optional cohort of 120 MBq, 4 to 6 cycles every 2 weeks
  Dose Level 3a
  - 160 MBq, 4 to 6 cycles every 4 weeks
  Dose Level 3b
  - Optional cohort of 160 MBq, 4 to 6 cycles every 2 weeks
  Dose Level 3c
  - Optional cohort of 160 MBq, 4 to 6 cycles every week
  Dose Level 4a
  * 200 MBq, 4 to 6 cycles every 4 weeks
  Dose Level 4b
  - Optional cohort of 200 MBq, 4 to 6 cycles every 2 weeks
  Dose Level 4c
  - Optional cohort of 200MBq, 4 to 6 cycles every week
  Ph2a Expansion
  Drug: [²¹²Pb]Pb-ADVC001 at recommended phase 2 dose and schedule

SUMMARY:
This is a prospective, open-label, non-randomised, dose-escalation and expansion study. The study aims to determine the safety and tolerability of escalating doses of [212Pb]Pb-ADVC001 administered every 6, 4, 2 or 1 week(s) during the dose finding phase (Phase 1b), and then aims to assess the efficacy and safety of [212Pb]Pb-ADVC001 at the RP2D in 3 participant groups in the expansion phase (Phase 2a).

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent for the trial.
* Adults aged 18 years or older at the time of consent.
* Has documented metastatic adenocarcinoma of the prostate, confirmed by histopathology.
* Has metastatic disease (≥ 1 metastatic lesion present on screening CT, magnetic resonance imaging [MRI] or bone scintigraphy scan).
* Has castration-resistant prostate cancer progressing or has progressed on androgen receptor therapy with castrate level of serum/plasma testosterone (≤ 50 ng/dL or ≤ 1.7 nmol/L). Progression at screening demonstrated by at least one of the following:

  1. Increase in PSA greater than 25% and > 2 ng/mL above nadir, confirmed by progression at two timepoints at least three weeks apart
  2. Progressive disease or new lesion(s) (relative to previous imaging) in the viscera or lymph nodes as per the Response Evaluation Criteria in Solid Tumours (RECIST) 1.1 or in bone as per Prostate Cancer Clinical Trials Working Group 3 (PCWG3). Any ambiguous results are to be confirmed by additional imaging modality (e.g., CT or MRI, Tc99m bone scintigraphy).
* For Phase 1b Dose Escalation: Exposure to at least one ARPi and taxane-based chemotherapy at any time in the course of their disease (unless taxanes considered contraindicated or declined by participant as documented in the patient's source documents and eCRF).
* For Phase 2a Expansion Group 1: Has had exposure to at least one ARPi at any time in the course of their disease.Has received at least one line of taxane-based chemotherapy for the treatment of mCRPC. Has not had exposure to ¹⁷⁷Lu-PSMA.
* For Phase 2a Expansion Group 2: Has had exposure to at least one ARPi at any time in the course of their disease. Has not received a taxane for the treatment of mCRPC. Note, participants may have received a taxane-based therapy in the (neo)adjuvant or mHSPC setting at least 12 months prior to C1D1. Has not had exposure to ¹⁷⁷Lu-PSMA.
* For Phase 2a Expansion Group 3: Has had exposure to at least one ARPi at any time in the course of their disease. Has had exposure to 177Lu-PSMA at any time in the course of their disease.
* Has disease that is prostate specific membrane antigen (PSMA) positive, as demonstrated by ⁶⁸Ga-PSMA-PET/CT or ¹⁸F-based PSMA PET/CT and confirmed as eligible by local reader. PSMA-positive participants are defined as those having at least one tumour lesion with ⁶⁸Ga- or ¹⁸F- PSMA PET CT uptake greater than normal liver (based on visual assessment) and all tumour lesions larger than size criteria with ⁶⁸Ga- or ¹⁸F-PSMA uptake greater than liver [short axis size criteria: organs ≥ 1 cm, lymph nodes ≥ 2.5 cm, bones (soft tissue component) ≥ 1 cm].
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1.
* Has adequate haematological, renal, and liver function, as defined by safety laboratory results at Screening.
* Estimated life expectancy > 6 months.
* Has the capacity to understand the study and be willing and able to comply with all study requirements, including the timing and nature of all required assessments.
* Agrees to comply with the radiation protection guidelines (including hospital admissions and isolation, where relevant) that are applied by the treating institution.
* Agrees to practice adequate precautions to prevent pregnancy in a partner to avoid potential problems associated with radiation exposure to the unborn child.

Exclusion Criteria:

* Has prostate cancer with known significant sarcomatoid or spindle cell or neuroendocrine small cell components, as determined by the Investigator. Participants with minor sarcomatoid, spindle cell or neuroendocrine small cell prostate cancer, but otherwise PSMA-expressing disease, may be eligible at the discretion of the Investigator.
* Has symptomatic dry eye, symptomatic dry mouth, Sjogren's syndrome or other pathologies affecting salivary gland function.
* Has received prior systemic radioligand therapy. Note, prior radium-223 exposure is not exclusionary. Prior exposure to 177Lu-PSMA is required for Group 3 participants in Phase 2a Expansion, provided treatment ceased at least 12 weeks prior to C1D1.
* Has received systemic anti-cancer therapy and/or radiation therapy within four weeks of C1D1 or has received any investigational agent within four weeks of C1D1. Note, patients should continue on androgen deprivation therapy. Prior ARPi therapy does not require washout prior to C1D1.
* Participants will not be eligible if any significant adverse events related to prior systemic anti-cancer therapy have not resolved to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE version 5.0) Grade ≤ 2 at the time of Screening, even if the systemic therapy ceased greater than four weeks prior to C1D1.
* Has malignancies other than prostate cancer within 3 years prior to enrolment, except for those with a negligible risk of metastases (e.g expected 5-year-overall-survival >90%) treated with expected curative outcome.
* Has known CNS metastases of any size.
* Has symptoms of spinal cord compression or impending spinal cord compression. Patients with prior treatment for spinal cord compression should be clinically stable off steroids for at least 4 weeks.
* Has diffuse bone-marrow involvement, i.e, "superscan", defined as bone scintigraphy in which there is excessive skeletal radioisotope uptake (>20 bone lesions) in relation to soft tissues, along with absent or faint activity in the genitourinary tract due to diffuse bone/bone marrow metastases).
* Has a serious active or sub-clinical infection, or angina pectoris, or heart failure (New York Heart Association [NYHA] Class III or IV), or significantly prolonged QT interval, or other serious illness which might impair the ability to participate in this study to the full extent, or which may require treatment that could interact with study treatment. Evidence of untreated urinary tract obstruction (e.g., hydroureter or hydronephrosis). Participants who undergo a successful decompressive procedure prior to treatment and participants with chronic, stable mild to moderate hydronephrosis without renal impairment will not be excluded.
* Has a known alteration in breast cancer genes (BRCA) BRCA1 or BRCA2 and are eligible to receive poly ADP ribose polymerase (PARP) inhibitor therapy according to their treating institution's standard of care. Note, participants with BRCA mutations who had disease progression on PARP inhibitors or who are not eligible for treatment with PARP inhibitors, are eligible.
* Has severe claustrophobia or other condition (e.g., pain) that may impact the ability to comply with the imaging aspects of this protocol.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
RP2D | Up to 60 Months
  Incidence and severity of dose-limiting toxicities, as defined in Section 6.5 of the protocol and assessed in accordance with NCI CTCAE Version 5.0.
  Incidence and severity of AEs and SAEs, assessed in accordance with NCI CTCAE Version 5.0.

SECONDARY OUTCOMES:
Maximum tolerated dose (MTD) | Up to 60 months
  Incidence and severity of dose-limiting toxicities, as defined in Section 6.5 of the protocol and assessed in accordance with NCI CTCAE Version 5.0.
Safety and Tolerability | Up to 60 months
  Incidence and severity of AEs and SAEs, assessed in accordance with NCI CTCAE Version 5.0.
Dosimetry | Day 1 of the first cycle through to the end of treatment (28 days after administration of the last treatment cycle).
  Absorbed radiation doses (expressed as Gy/MBq) of administered [²¹²Pb]Pb-ADVC001 to organs at risk and tumour lesions.
Preliminary therapeutic efficacy as assessed by PSA response | Up to 60 months
  PSA response defined as a reduction from baseline PSA level of at least 50% (PSA 50) and 90% (PSA 90), confirmed by a follow-up PSA.
Preliminary therapeutic efficacy as assessed by objective response rate and disease control rate | Up to 60 months
  Objective response rate (OCR) and disease control rate (DCR) derived from CT imaging based on RECIST 1.1 and Prostate Cancer Trials Working Group 3.
Preliminary therapeutic efficacy as assessed by radiographic progression-free survival | Up to 60 months
  Radiographic progression-free survival (rPFS) defined as the time from date of first dosing to the occurrence of one of the following:
  1. Progression of measurable lesions using RECIST 1.1.
  2. Progression of bone lesions using Prostate Cancer Working Group 3 criteria.
  3. Death due to any cause.
Preliminary therapeutic efficacy as assessed by progression-free survival | Up to 60 months
  Progression-free survival defined as the time from date of first dosing to the occurrence of one of the following:
  1. Radiographic progression per RECIST 1.1 or bone scan in accordance with PCWG3 criteria.
  2. Clinical progression as determined by investigator assessment.
  3. PSA progression defined by PCWG3.
  4. Death due to any cause.
Preliminary therapeutic efficacy as assessed by overall survival | Up to 60 months
  Overall survival defined as the time from date of first dosing to death from any cause.

OTHER OUTCOMES:
Biodistribution | Up to 24 weeks
  Biodistribution of [²¹²Pb]Pb-ADVC001 on SPECT/CT and [⁶⁸Ga]Ga-PSMA (or [¹⁸F]F-based-PSMA) on PET/CT as determined by image analysis and interpretation by expert readers.
PSMA PET response | Up to 24 weeks
  [⁶⁸Ga]Ga- or [¹⁸F]F-based PSMA responses based on the Consensus Statement on PSMA PET Response Assessment Criteria in Prostate Cancer.
Biomarkers of immune activation | Up to 32 weeks
  Change from baseline in biomarkers of immune activation and efficacy endpoints including PSA response and ORR.
PK parameter: Maximum observed concentration (Cₘₐₓ) of [²¹²Pb]Pb-ADVC001 | On the first and second day of study treatment
PK parameter: Time to maximum observed concentration (Tₘₐₓ) of [²¹²Pb]Pb-ADVC001 | On the first and second day of study treatment
PK parameter: Area under the concentration-time curve (AUC) of [²¹²Pb]Pb-ADVC001 | On the first and second day of study treatment
PK parameter: Clearance of [²¹²Pb]Pb-ADVC001 | On the first and second day of study treatment
Exploratory [²¹²Pb]Pb PET/CT imaging | Up to 5 weeks
  Biodistribution of [²¹²Pb]Pb-ADVC001 via [²¹²Pb]Pb PET/CT.
Patient Reported Outcomes (PRO) | Up to 32 weeks
  Change from baseline in "Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events" scores, where responses range from "Never," "Not at all," and "None" at their best to "Almost constantly," "Very much," and "Very severe" at their worst.

CONTACTS AND LOCATIONS:
Overall Officials: David Wyld, Principal Investigator — Royal Brisbane & Women's Hospital; Aaron Hansen, Principal Investigator — Princess Alexandra Hospital
Locations (2):
- Australia (2):
  - Royal Brisbane & Women's Hospital, Brisbane, Queensland
  - Princess Alexandra Hospital, Brisbane, Queensland

IPD SHARING:
Plan to Share IPD: No